CLINICAL TRIAL: NCT04783636
Title: A Randomized, Open-label, Single-dosing, 2x2 Crossover Phase 1 Study to Compare the Safety and Pharmacokinetics of PT105 With PT105R in Healthy Postmenopausal Female Volunteers
Brief Title: To Compare the Safety and Pharmacokinetics of PT105 With PT105R in Healthy Postmenopausal Female Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peptron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PT105-BE
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Other): After a single administration of PT105R (leuprorelin acetate 3.75mg), a single administration of PT105 (leuprorelin acetate 3.75mg)
  Interventions: Drug: leuprorelin acetate 3.75mg
- B (Other): After a single administration of PT105 (leuprorelin acetate 3.75mg), a single administration of PT105R (leuprorelin acetate 3.75mg)
  Interventions: Drug: leuprorelin acetate 3.75mg

INTERVENTIONS:
Drug: leuprorelin acetate 3.75mg — PT105, PT105R
  Other Names: PT105

SUMMARY:
The purpose of study is to compare the safety and pharmacokinetics of PT105 with PT105R in healthy postmenopausal female volunteers

DETAILED DESCRIPTION:
The purpose of study is to confirm the safety and pharmacokinetics of PT105 in healthy postmenopausal female volunteers

ELIGIBILITY:
Inclusion Criteria:

* A healthy woman who is over 19 years of age and has been certified obstetrically with menopause, at the time of screening.
* Subjects weighing over 50 kg with BMI between 18 and 30 kg/m2 (inclusive) at screening visit.

Exclusion Criteria:

* Those who have clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history
* Those whose plasma AST and ALT exceed 2 times to the upper limit of the normal range in screening including additional examinations prior to randomization
* Subjects who have participated and taken investigational drug in any other clinical trial (including bioequivalence study) within six months prior to study drug administration
* Subjects who have donated a unit of whole blood within two months or blood components within one month prior to study drug administration

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-11 (Estimated); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-07-20 (Estimated)

PRIMARY OUTCOMES:
AUC7-t of Leuprolide | 0h, 0.5, 1, 2, 4, 8, 12, 24, 72, 168, 240, 336, 504, 672, 840, 1008 hr
  AUC7-t
AUCt of Leuprolide | 0h, 0.5, 1, 2, 4, 8, 12, 24, 72, 168, 240, 336, 504, 672, 840, 1008 hr
  AUCt
AUCinf of Leuprolide | 0h, 0.5, 1, 2, 4, 8, 12, 24, 72, 168, 240, 336, 504, 672, 840, 1008 hr
  AUCinf
Cmax of Leuprolide | 0h, 0.5, 1, 2, 4, 8, 12, 24, 72, 168, 240, 336, 504, 672, 840, 1008 hr
  Cmax

SECONDARY OUTCOMES:
Tmax of Leuprolide | 0h, 0.5, 1, 2, 4, 8, 12, 24, 72, 168, 240, 336, 504, 672, 840, 1008 hr
  Tmax
t1/2 of Leuprolide | 0h, 0.5, 1, 2, 4, 8, 12, 24, 72, 168, 240, 336, 504, 672, 840, 1008 hr
  t1/2

IPD SHARING:
Plan to Share IPD: No